CLINICAL TRIAL: NCT04046471
Title: Weight Management for Adults With Mobility Related Disabilities
Brief Title: Weight Loss Physical Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 142753; 1R01DK116669-01A1 (NIH)
Record Dates: First submitted 2019-07-31; First posted 2019-08-06 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Physical Disability
Keywords: Weight Loss; Physical Activity; Diet
MeSH Terms: conditions — Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual In-Person (Other)
  Interventions: Dietary Supplement: enhanced Stop Light Diet; Behavioral: Individual In-Person
- Group Remote (Other)
  Interventions: Dietary Supplement: enhanced Stop Light Diet; Behavioral: Group Remote

INTERVENTIONS:
Dietary Supplement: enhanced Stop Light Diet — Stop light diet enhanced with portion-controlled meals
Behavioral: Group Remote — Participants will receive remotely delivered weight loss in a group setting.
  Arms: Group Remote
Behavioral: Individual In-Person — Participants will receive a weight loss intervention during individual, at-home visits.
  Arms: Individual In-Person

SUMMARY:
The objective of this study is to compare weight loss (6 mos.) and maintenance (18 mos.) between an individual home visit intervention (IH) and an intervention delivered remotely via video conferencing to groups of overweight/obese adults with Mobility Related Disabilities (MRDs) in their homes (GR). The primary aim will be to compare weight loss (0-6 mos.) between the two interventions (IH vs. GR). Secondarily, the study team will compare the mean weight loss from 0-18 mos., the proportion of participants achieving >=5% weight loss from baseline, changes in cardiovascular risk factors and quality of life, and conduct a cost analysis. In addition, factors that will be explored include the influence of behavioral session attendance, compliance with the recommendations for diet (energy intake, number of entrees/shakes, servings of fruits/vegetables), Physical Activity (PA, min of moderate vigorous PA, min sedentary time), and self-monitoring of diet and PA, self-efficacy for dietary change and PA, dietary self-regulation, social support for diet/PA, barriers to PA, sleep and medications on weight loss at 6 and 18 mos.

DETAILED DESCRIPTION:
The investigators propose a 2-arm randomized trial (group remote (GR) vs. individual home visit (IH)) using intent-to-treat principles, to compare body weight following weight loss (6 mos.) and maintenance (18 mos.) in overweight/obese adults with Mobility Related Disabilities (MRDs). Adults with MRDs (n=128) will be randomized (1:1) to one of the 2 intervention arms for an 18-mo. trial (6 mos. weight loss, 12 mos. maintenance). Cohorts of ~30-45 individuals will be recruited. Following baseline testing, participants will be stratified by their primary mode of locomotion outside the home, i.e., ambulatory or assistive device (wheelchair, scooter, etc.), and randomized with equal allocation to GR or IH arms. Both interventions will be delivered in a format that eliminates the transportation barrier, prescribed an enhanced stop light diet, and will self-monitor body weight using electronic scales. The GR arm will include group behavioral counseling and group PA delivered remotely via video conferencing (Zoom trademark software) on a tablet computer (iPad mini) to participants in their homes, and use commercially available web-based applications for self-monitoring/participant feedback for diet (Lose It! software) and PA (Fitbit activity tracker). The IH arm will include behavioral counseling delivered during individual home visits, a prescription for self-directed PA, and self-monitoring of diet and PA using conventional paper and pencil self-reports. All outcomes will be collected by trained research assistants who are blinded to the study condition. The primary aim will be to compare weight loss (0-6 mos.) between the GR and IH interventions. Secondarily, the research team will compare mean weight loss from 0-18 mos., the proportion of participants achieving >=5% weight loss from baseline, changes in cardiovascular risk factors and quality of life, and conduct a cost analysis. In addition, the influence of behavioral session attendance, compliance with the recommendations for diet (energy intake, number of entrees/shakes, servings of fruits/vegetables), PA (min of moderate-vigorous PA, min sedentary time), and self-monitoring of diet and PA, self-efficacy for dietary change and PA, dietary self-regulation, social support for diet/PA, barriers to PA, sleep, and medications on weight loss between the IH and GR arms will be explored, with 80% power and a type 1 error rate of 0.05, assuming a common standard deviation of 6 kg, will require 64 participants/group. A 2-sample independent t-test will be used to compare 6 mo. weight loss (primary aim) between the 2 intervention arms in both an intent-to-treat and completer only analysis. For the secondary aim 1, comparison of 18 mo. weight loss, will mirror the analysis for the primary aim. A 2-sample t-test will be used to compare weight change (0-18 mos.) between the 2 intervention arms. For secondary aim 2, a between arm comparison of the proportion of participants achieving >=5% weight loss (0-18 mos.) will be evaluated using a chi-square test. Secondary aims 3 and 4, between arm comparison of change in risk factors and quality of life (0-6 and 0-18 mos.), will be evaluated using a 2-sample ttest. Exploratory aims will examine the influence of the following on weight loss at 6 mos.: behavioral session attendance; compliance with the recommendations for diet (energy intake, number of entrees/shakes, servings of fruits/vegetables), PA (min of moderate-vigorous PA, min sedentary time), self-monitoring of diet and PA, sleep, and medications assessed over the time period of interest i.e. (0-6 and 0-18 mos.); and the changes in self-efficacy for PA and dietary change, dietary self-regulation, social support for diet/PA, and barriers to PA from 0-6 mos. The influence of these factors as covariates will be examined, in addition to treatment, on weight loss at 6 mos. This will allow the ability to identify which variables most highly influence the outcome along with treatment and/or the mechanism(s) of action that are impacting weight loss.

ELIGIBILITY:
Inclusion Criteria:

* A permanent MRD (>= 1 yr. duration) requiring the use of a wheelchair or resulting in the inability to walk 0.25 miles without stopping, with or without assistive devices, as documented by 7 items from the NHANES Physical Funding Survey (113), and confirmed by the Primary Care Physician (PCP). Individuals with MRDs, associated with, but not limited to spinal cord injury (SCI), spina bifida, multiple sclerosis, cerebral palsy, stroke, muscular dystrophy, and lower limb amputation will be included.
* Age 18 yrs and above. Weight management for younger individuals requires different behavioral strategies.
* Body mass index (BMI) above 25 kg/m squared. Individuals with BMI, with a BMI <25kg/m squared are not overweight. We are aware of the difficulty in the assessment of BMI, and issues related to the use of BMI for classifying overweight/obesity in individuals with SCI or amputations. Thus, in questionable cases we will defer to the PCP regarding eligibility based on weight status.
* Wireless internet access in the home.

Exclusion Criteria:

* Unable to participate in light-to-moderate intensity PA, e.g., seated aerobics, resistance exercise, or physically unable to use the iPad.
* Participation in a structured weight loss or exercise program in the previous 6 mos. These proximal exercises may influence this trial.
* Not weight stable (plus/minus 4.6 kg) for 3 mos. prior to intake.
* Unwilling to be randomized.
* Pregnancy during the previous 6 mos. currently lactating, or planned pregnancy in the following 18 mos.
* Serious medical risk, e.g., cancer, recent heart attack, stroke as determined by the PCP.
* Current use of antipsychotics, untreated depression, or other psychiatric illness that would preclude participation in weight management, as determined by the PCP. Psychiatric co-morbidity may limit the benefits from health education. Addressing psychiatric issues is beyond the scope of this study.
* Cognitive, visual, or hearing impairments that may interfere with compliance to the study protocol as determined by the PCP.
* Adherence to specialized diets, e.g., food allergies, vegetarian, macrobiotic.
* Binge (Binge Eating Scale) or other eating disorders (EATs-26).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Donnelly, EdD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Washburn RA, Ptomey LT, Gorczyca AM, Smith PR, Mayo MS, Lee R, Donnelly JE. Weight management for adults with mobility related disabilities: Rationale and design for an 18-month randomized trial. Contemp Clin Trials. 2020 Sep;96:106098. doi: 10.1016/j.cct.2020.106098. Epub 2020 Aug 6. PMID 32768682

RESULTS

PARTICIPANT FLOW:
Period: 6-month
Arm/Group | Individual In-Person | Group Remote
Started | 63 | 66
Completed | 54 | 62
Not Completed | 9 | 4
Period: 12-month
Arm/Group | Individual In-Person | Group Remote
Started | 54 | 62
Completed | 49 | 58
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual In-Person | Group Remote | Total
Number analyzed (Participants) | 63 | 66 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 42 | 90
  >=65 years | 15 | 24 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12.4) | 55.9 (14.3) | 55.1 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 53 | 103
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 53 | 58 | 111
  Unknown or Not Reported | 9 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 6 | 16
  White | 45 | 55 | 100
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 63 | 66 | 129

OUTCOME MEASURES:

1. Primary Outcome: Weight Change in kg From Baseline to 6-months
Description: Weight will be measured in duplicate with a portable, calibrated digital scale. (Model #PS6600, Befour, Saukville, WI.). For those in a wheelchair, weight will be measured in duplicate using a portable calibrated, digital wheelchair scale (Model MX420, Befour, Saukville, WI.). Participant weight will be calculated as participant + chair weight minus chair weight.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Individual In-Person | Group Remote
Number analyzed (Participants) | 63 | 66
kg | -6.23 (6.70) | -8.16 (6.74)

2. Secondary Outcome: Weight
Description: as for outcome 1
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

3. Secondary Outcome: Waist Circumference
Description: Measured in cm around narrowest part of the waist.
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

4. Secondary Outcome: Blood Pressure
Description: Obtained with an automated sphygmomanometer (DinaMap ProCare 100, General Electric) using the NHANES blood pressure protocol.
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Quality of Life
Description: Assessed with the SF-36E. The SF-36E measures quality of life on a 0-100 scale with 0 being low quality and 100 being high quality.
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

6. Secondary Outcome: Cost of Intervention
Description: The cost of both the IH and GR interventions will be calculated along with the cost per additional kg of weight loss.
Time Frame: Across 18 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Compliance With the Diet Recommendations
Description: Will be assessed using photo-assisted food records over 4 consecutive days (3 wk. days and 1 wk. end day) starting the weekend prior to scheduled outcome assessments.
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Compliance With Physical Activity Recommendations
Description: Assessed using the Physical Activity and Disability Survey (PADS). The PADS is a semi-structured interview that includes subscales for exercise, leisure time PA, household activity, and inactivity (sleeping, TV, computer use).
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Behavioral Session Attendance
Description: Expressed as the percentage of possible sessions attended
Time Frame: Across 18 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Self-monitoring of Diet/PA
Description: The percentage of prescribed monitoring days completed across 18 mos.
Time Frame: Across 18 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Self-efficacy for Dietary Change
Description: Assessed using the Weight Efficacy Lifestyle Scale. This scale has participants rate a question from 1 to 10 with 1 being "Not at all confident" and 10 being "Very confident."
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Barriers to Exercise
Description: Assessed using the Barriers to Exercise for Disabled Person. Individuals are asked a question relating to a specific exercise barrier and if it has limited their participation in the past three months. If they answer yes, they are asked to rate the limitation of that barrier on a scale of 1 to 5 with 1 being the least and 5 being the most limiting. Scores are calculated using weighted sums of the items.
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Diet Self-regulation
Description: Assessed using the Three-Factor Eating Inventory, a widely-used measure of eating behavior (restraint, disinhibition, hunger). Participant is asked a question and to rate how they feel on a 1-4 scale with 1 being "definitely false" and 4 being "definitely true."
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Social Support
Description: Social support for both exercise and dietary habits will be assessed using the Social Support and Exercise/Diet Survey. This survey utilizes questions focusing on support by peers and family members that participants answer using a 1-5 rating with 1 being "no support" and 5 being "very supportive."
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Sleep
Description: Sleep Quality will be assessed using The Pittsburgh Sleep Quality Index. Participants answer open-ended questions as well as questions on a 0-3 scale. Seven component scores are tallied using provided measures, and a global sum of "5"or greater on all seven components indicates a "poor" sleeper.
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Medication Information
Description: Medication name/frequency/amount will be collected by participant self-report
Time Frame: Baseline, 6, 12, and 18 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Energy Expenditure
Description: Energy expenditure of the remote sessions will be assessed in a volunteer sample using a previously validated portable, open-circuit indirect calorimeter (Cosmed, Italy) which measures breath-by-breath ventilation, expired oxygen, and carbon dioxide.
Time Frame: 3-12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to 6-months
Arm/Group | Individual In-Person | Group Remote
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/66
Serious Adverse Events (participants affected / at risk) | 4/63 | 2/66
Other Adverse Events (participants affected / at risk) | 0/63 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individual In-Person (N=63) | Group Remote (N=66)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lupus Flare (Immune system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Smoke Inhalation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Heart Failure Complications (General disorders) | 1 (1) | 0 (0)
Aortic Stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Bladder Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT04046471/Prot_SAP_000.pdf